CLINICAL TRIAL: NCT01504282
Title: Mitomycin-c Application for Photorefractive Keratectomy
Brief Title: Mitomycin-c Application for PRK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 8901
Record Dates: First submitted 2012-01-04; First posted 2012-01-05 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2010-06

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Mitomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- MMC group (Active Comparator): One eye of each patient was randomly assigned to receive intraoperative topical 0.02% MMC for 5 seconds.
  Interventions: Drug: mitomycin-C
- BSS group (Placebo Comparator): One eye of each patient was randomly assigned to receive balanced salt solution (BSS) with the same manner.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: mitomycin-C
  Arms: MMC group
Drug: Placebo — balanced salt solution (BSS)
  Arms: BSS group

SUMMARY:
To evaluate the safety and efficacy of 5 seconds mitomycin-C (MMC) application during photorefractive keratectomy (PRK) for patients with low myopia.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria was ablation depth less than 65 µm,
* a stable refractive error for at least 1 year
* corrected distance visual acuity (CDVA) of 0.1 LogMAR or better.

Exclusion Criteria:

* Patients with keratoconus suspect,
* excessive dry eyes,
* impaired wound healing processes,
* lenticular changes,
* corneal dystrophy,
* history of ocular surgery,
* anterior or posterior uveitis,
* glaucoma and retinal diseases were excluded.

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 90

PRIMARY OUTCOMES:
Central corneal endothelial cell density (ECD) 6 months after the PRK | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Tehran Province, Iran